CLINICAL TRIAL: NCT00700674
Title: Is the Ese of EEG Entropy as Intra-operative Monitor Improves Postoperative Cognitive Dysfunction
Brief Title: Effect of Usage of Electroencephalogram (EEG) Entropy on the Incidence of Postoperative Cognitive Dysfunction in Geriatric Patients
Status: Terminated | Type: Observational
Why Stopped: Progress report requested by Dr. Abboud decided to close it.
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: RP 0729
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2010-02

CONDITIONS: Cognitive Dysfunction
Keywords: EEG entropy; Elderly; Decreases; POCD; Use of EEG entropy; Geriatric
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Entropy group
- 2: Control

SUMMARY:
To determine if the usage of EEG Entropy helps to reduces the incidence of POCD in elderly patients after general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II.
* scheduled for retinal surgery expected to take 2-3 hours under general anesthesia.
* orotracheal intubation.

Exclusion Criteria:

* history of cardiac, pulmonary, liver or renal disease.
* significant obesity (body mass index >30.
* Long-term user of central nervous system activator drugs, benzodiazepines and/or opiates.
* dementia, brain atrophy and other neurological disorder.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 Elderly patient, ASA 1-2
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Riad, MD,AB,SB, Principal Investigator — King Khaled Eye Specialist Hospital
Locations (1):
- King Khaled Eye Specialist hospital, Riyadh, Saudi Arabia